CLINICAL TRIAL: NCT00213187
Title: The Effect of Vigorous Exercise on Motor Function and Functional Fitness in Juvenile Arthritis
Brief Title: PEAK Study (Physical Exercise and Activity in Kids)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Rheumatology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0020020201; 137845 (CIHR)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile Rheumatoid Arthritis,; Randomized Control Trial,; attention placebo,; exercise testing,; aerobics,; Qi Gong,; exercise video,; activities of daily living,; quality of life,; economy of walking,; fitness; pediatrics
MeSH Terms: conditions — Arthritis, Juvenile

INTERVENTIONS:
Behavioral: Aerobic and Qi gong Exercise

SUMMARY:
The objectives of this study are to study the effect of formal exercise training on motor function and overall physical fitness in children with arthritis. A 12-week comprehensive exercise program will be used. Formal exercise training will be compared to Qi gong.

DETAILED DESCRIPTION:
Childhood arthritis is a common and often debilitating disease. Children with arthritis are less active than their peers, and consequently they often have poor physical fitness. This study follows up our pilot study, in which we showed that exercise training can be safely carried out in children who have arthritis.

We plan to randomly assign 80 children with arthritis to one of two groups. The experimental group undergoes a vigorous exercise training program consisting of twelve weekly supervised sessions as well as twice weekly at home sessions using an exercise video. The control group also has twelve supervised sessions and two home sessions. However, their exercises are non-strenuous, based on Qi gong. All children have comprehensive fitness testing before and after the training at the exercise lab at the Hospital for Sick Children.

If we show that fitness exercise leads to improved motor function and improved ability to carry out activities of daily living, then we will change the way in which we provide therapy for childhood arthritis. We hope that this study will lead to an improved quality of life for children with arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 - 16 years.
2. Diagnosis of Juvenile Idiopathic Arthritis - based on the revised Durban criteria.
3. Polyarticular or pauciarticular course.
4. Stable Disease - on a stable dose of NSAID, and if applicable methotrexate or other second line agents - in the preceding month, and judged by the attending rheumatologist to be clinically stable and unlikely to need a change in medication over the course of the trial.
5. Medications. There are no restrictions on medication use for this study; however, every effort is made to keep medication dosage stable over the course of study.

Exclusion Criteria:

1. Co-morbidity with cardiac, pulmonary or metabolic disease.
2. Moderate or severe hip pain while walking (as judged by the patient and scored on a 4 point scale) or active systemic symptoms (fever, rash).
3. Children who engage in more than 3 hours of structured extracurricular physical activity weekly may not show additional gains from fitness training and, therefore, are not studied. Children are not otherwise excluded from the study if currently attending a physiotherapy pool program with emphasis on joint range of motion and stretching.
4. Children who are unable to cooperate with testing procedures.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80
Dates: Start 2002-08; Study Completion 2005-11

PRIMARY OUTCOMES:
walking economy at completion of the exercise program
PEAK power, muscular endurance, and subjective function at completion of the exercise program

SECONDARY OUTCOMES:
Peak aerobic capacity (VO2 peak) measured post-exercise program
Anaerobic Power as measured by a Modified Wingate test at completion of the exercise program
Anthropometry as measured by Body Mass Index (BMI) and skinfold at completion of the exercise program
Improved physical function measured post treatment
Improved daily activity measured post treatment
Improved quality of life measure post treatment
Decreased arthritis activity measured post treatment
Improved range of motion measure post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brian M. Feldman, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Stephens S, Singh-Grewal D, Bar-Or O, Beyene J, Cameron B, Leblanc CM, Schneider R, Schneiderman-Walker J, Selvadurai H, Silverman E, Spiegel L, Tse SM, Wright V, Feldman BM. Reliability of exercise testing and functional activity questionnaires in children with juvenile arthritis. Arthritis Rheum. 2007 Dec 15;57(8):1446-52. doi: 10.1002/art.23089. PMID 18050186
- [Derived] Singh-Grewal D, Schneiderman-Walker J, Wright V, Bar-Or O, Beyene J, Selvadurai H, Cameron B, Laxer RM, Schneider R, Silverman ED, Spiegel L, Tse S, Leblanc C, Wong J, Stephens S, Feldman BM. The effects of vigorous exercise training on physical function in children with arthritis: a randomized, controlled, single-blinded trial. Arthritis Rheum. 2007 Oct 15;57(7):1202-10. doi: 10.1002/art.23008. PMID 17907238